CLINICAL TRIAL: NCT05636462
Title: Effects of Global Postural Re-education Program on Neck Pain and Disability in Breast Feeding Females.
Brief Title: Global Postural Re-education Program on Neck Pain in Breast Feeding Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Feryal Arshad
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain; Disability Physical; Breast Feeding
MeSH Terms: conditions — Neck Pain; Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global postural re-education (Experimental): It consists of 27 patients who will receive conventional exercises and global postural re-education which will be divided in three components First in lying posture to stretch anterior muscles of neck for 15 min, second component in supine position and stretching posterior muscles for 15 min and final component is in standing position under a load of gravity for 5 min for 3 days a week .
  Interventions: Other: Global postural re-education program
- Conventional Physical therapy (Active Comparator): It consists of 27 patients who will receive conventional therapy including stretching and strengthening exercises of neck for 3 days a week.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Global postural re-education program — Different postures of global re-education programs are used and stretch is applied in these postures.
  3 sessions per week are given and each session time is 40 minutes. Treatment is given for 4 weeks.
  Arms: Global postural re-education
Other: Conventional Physical Therapy — Isometrics and stretching is used as conventional treatment. 3 sessions per week are given and each session time is 40 minutes. Treatment is given for 4 weeks.
  Arms: Conventional Physical therapy

SUMMARY:
The significance of this study is that it will add to the growing body of knowledge that if these techniques yield outcomes in treatment of neck pain in breast feeding mothers. This study will add the beneficial effects to treat the neck pain in breast feeding females.

DETAILED DESCRIPTION:
Nonspecific neck pain is an increasingly frequent musculoskeletal condition affecting 22% to 70% of the population that is more prevalent in women than in men. Some patients will not experience complete resolution of pain and disability which can become a more complex chronic pain syndrome.(2) When symptoms persist for more than 12 weeks, the condition acquires the value of chronicity and is denominated chronic nonspecific neck pain. This is associated with high costs for public health, and is becoming a socio-health problem.

The mechanisms underlying recurrence or persistence of neck pain may be associated with biomechanical, functional, proprioceptive, and postural changes. However, the multidimensional nature of neck pain can involve not only the sensory-motor component, but also psychosocial components, such as anxiety, depression, and fear and catastrophic thoughts in response to pain (kinesiophobia and pain catastrophizing).

In 2018, a study is conducted on the effect of global postural reeducation in patients with chronic nonspecific neck pain and their study suggested that global postural reeducation shows promising results for the improvement of neck pain and disability in patients with chronic neck pain.

In 2016, a randomized controlled trial is conducted on Effectiveness of Global Postural Re-education in Patients With Chronic Nonspecific Neck Pain The result of the study showed that global postural reeducation , when provided in the absence of other intervention, can significantly decrease pain Pain intensity , disability and increases cervical range of motion.

In 2015, a research is conducted to find out the effects in short and long term of global postural reeducation (GPR) on chronic low back pain the result showed that global postural reeducation is effective in the treatment of low back pain and function this study, suggests that postural reeducation was highly effective in managing pain and function due to low back.

Although quite a number of researches have been done regarding more effective treatment of neck pain, there are actually no research in effect of postural re-education is seen in breast feeding females.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-35 Years
* Mothers who have pain score of 4 in NPRS
* Mothers who breast feed their babies
* Post-partum period

Exclusion Criteria:

* Neck pain due to any other comorbidity e.g. Previous history of trauma or fracture, disc prolapse, facet joint stenosis
* Previously kyhoscoliotic mothers
* Females who have C-section

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Neck pain | 4th day
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a uni dimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases. Validity 0.86 to 0.95
Neck Disability Index | 4th day
  The most used neck disability questionnaires are the Neck Pain and Disability scale (NPAD) and the Neck Disability Index (NDI) The Neck Pain and Disability scale (NPAD) is a composite index including 20 items which measure the intensity of neck pain and related disability,reliability between 0,50 and 0,98

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, Mphil, Principal Investigator — Riphah International University
Locations (1):
- PSRD, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendes-Fernandes T, Puente-Gonzalez AS, Marquez-Vera MA, Vila-Cha C, Mendez-Sanchez R. Effects of Global Postural Reeducation versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women with Chronic Nonspecific Neck Pain: Study Protocol for a Randomized, Parallel, Clinical Trial. Int J Environ Res Public Health. 2021 Oct 12;18(20):10704. doi: 10.3390/ijerph182010704. PMID 34682453
- [Background] Somarajan S, Hingarajia D. Effect of Global Postural Re-Education and Static Stretching on Pain and Disability in Women with Chronic Non-Specific Neck Pain-A Comparative Study. Indian Journal of Public Health Research & Development. 2021;12
- [Background] Cavalcanti IF, Antonino GB, Monte-Silva KKD, Guerino MR, Ferreira APL, das Gracas Rodrigues de Araujo M. Global Postural Re-education in non-specific neck and low back pain treatment: A pilot study. J Back Musculoskelet Rehabil. 2020;33(5):823-828. doi: 10.3233/BMR-181371. PMID 31929138